CLINICAL TRIAL: NCT01719744
Title: A Phase II Study of Oral ENMD-2076 Administered to Patients With Advanced/Metastatic Soft Tissue Sarcoma
Brief Title: Study of ENMD-2076 in Patients With Advanced/Metastatic Soft Tissue Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2076-STS-001
Record Dates: First submitted 2012-10-30; First posted 2012-11-01 (Estimated); Results first posted 2017-11-07 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Advanced; Metastatic; Soft Tissue Sarcoma
Keywords: ENMD-2076; advanced; metastatic; soft tissue sarcoma
MeSH Terms: conditions — Neoplasm Metastasis; Sarcoma | interventions — ENMD 2076

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ENMD-2076 (Experimental): ENMD-2076 capsules, 275 mg once daily, by mouth.
  Interventions: Drug: ENMD-2076

INTERVENTIONS:
Drug: ENMD-2076

SUMMARY:
This is a phase 2 study of ENMD-2076 in patients with advanced/metastatic soft tissue sarcoma. This study will help to understand how well ENMD-2076 works and how safe and tolerable the drug is in this patient population.

DETAILED DESCRIPTION:
ENMD-2076 is an oral drug that works by blocking certain enzymes called Aurora A from working. These enzymes are needed for cells to divide including cancer cells. ENMD-2076 also works by stopping the growth of new blood vessels which would provide the tumor with nutrients for it to grow. It is believed that by blocking Aurora A enzymes from working and stopping new blood vessels from growing, the tumors may stop growing or shrink.

ELIGIBILITY:
Inclusion Criteria:

* Have documented histological diagnosis of soft tissue sarcoma (e.g. leiomyosarcoma, synovial sarcoma, angiosarcoma and liposarcoma etc), with the exception of gastrointestinal stromal tumor (GIST).
* Meet revised RECIST criteria (version 1.1) within 4 weeks of entry by having measurable disease defined as one or more lesions that can be accurately measured in one or more dimensions. Areas of previous radiation may not serve as measurable disease unless there has been objective interval tumor growth documented radiologically.
* Must have had no more than 1 line of treatment in the advanced/metastatic setting. The use of prior anti-angiogenic therapy is allowed. Previous neo-adjuvant or adjuvant therapies are allowed.
* Are at least 3 weeks from major surgery or radiation therapy and recovered; 3 weeks from any other previous anticancer therapy and recovered including biologics.
* Are ≥ 18 years of age
* The patient has a multigated acquisition (MUGA) scan with an actual left ventricular ejection fraction of greater than or equal to the institution lower limit of normal within one month prior to start of study.
* Have clinically acceptable laboratory screening results within certain limits specified below:

  * AST and ALT ≤ 2.5 times upper limit of normal (ULN) or less than or equal to 5 times ULN if liver metastases are present
  * Total bilirubin ≤ 1.5 x ULN
  * Creatinine ≤ 1.5 x ULN or > 50 ml/min calculated by the Cockcroft and Gault formula (formula defined in appendix E).
  * Absolute neutrophil count ≥ 1500 cells/mm3
  * Platelets ≥ 100,000/mm3
  * Hemoglobin ≥ 9.0 g/dL
  * INR ≤ 1.5
* Have an ECOG performance status of 0 or 1.
* Patients must have and consent for access to archival material (for correlative studies). Patients who do not have archival material will be eligible if they consent for fresh tissue biopsy.
* Women of child producing potential must agree to use effective contraceptive methods prior to study entry, during study participation, and for at least 30 days after the last administration of study medication. A serum pregnancy test within 72 hours prior to the initiation of therapy will be required for women of childbearing potential.
* Have the ability to understand the requirements of the study, provide written informed consent which includes authorization for release of protected health information, abide by the study restrictions, and agree to return for the required assessments.
* Able to tolerate oral medications.

Exclusion Criteria:

* Women who are pregnant or nursing
* Have active, acute, or chronic clinically significant infections or bleeding.
* Have uncontrolled hypertension (systolic blood pressure greater than 150mmHg or diastolic blood pressure greater than 100mmHg); or history of congestive heart failure (equal to or greater than Grade 2 classification by New York Heath Association).
* Have active angina pectoris, stroke or recent myocardial infarction (within 6 months).
* Have chronic atrial fibrillation or QTc interval corrected for heart rate of greater than 480 msec.
* Have additional uncontrolled serious medical or psychiatric illness.
* Require therapeutic doses of anti-coagulation either by virtue of low-molecular weight heparin or coumadin (prophylactic anti-coagulation allowed). Patients with previous history of deep venous thrombosis or pulmonary embolism are also excluded.
* Known CNS metastases
* Have any medical condition that would impair the administration of oral agents including recurrent bowel obstructions, inflammatory bowel disease or uncontrolled nausea, vomiting or diarrhea
* Have 2+ protein by urinalysis. Patients with an ongoing or previous history of nephrotic syndrome will be excluded
* Have an additional malignancy diagnosed within 5 years of study enrollment with the exception of basal or squamous cell skin cancer or cervical cancer in situ
* Require treatment with drugs known to be potent inducers or inhibitors of CYP3A4 that cannot be substituted
* Patients who cannot or refuse to stop herbal medications of illicit drug use will be excluded from the study. Use of medical marijuana is not permissible in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-01; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Albiruni Razak, MBBS, Principal Investigator — Princess Margaret Cancer Centre
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- ENMD-2076: ENMD-2076 capsules, 275 mg once daily, by mouth.
  ENMD-2076
Period: Overall Study
Arm/Group | ENMD-2076
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | ENMD-2076
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 21
  >=65 years | 4
Age, Continuous [Median (Full Range); unit: years] | 54 [22 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 7
Region of Enrollment [Number; unit: participants]
  Canada | 25

OUTCOME MEASURES:

1. Primary Outcome: 6-month Progression-free Survival Rate (PFS)
Description: Number of patients with no progression of disease at 6 months
Time Frame: From start of study treatment until disease progression or death, whichever occurs first, up to 6 months.
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | ENMD-2076
Number analyzed (Participants) | 25
participants | 12 [3 to 31]

2. Secondary Outcome: Number of and Severity of Adverse Events Per Participant
Description: Number of participants who experienced a grade 3 or higher adverse event. Reporting threshold 5%
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | ENMD-2076
Number analyzed (Participants) | 25
participants
  HYPERTENSION | 16
  DIARRHEA | 4
  ALANINE AMINOTRANSFERASE INCREASED | 2
  ASPARTATE AMINOTRANSFERASE INCREASED | 2
  VOMITING | 2
  BLOOD BILIRUBIN INCREASED | 2
  HYPOKALEMIA | 2
  LUNG INFECTION | 2
  HYPOXIA | 2
  DEHYDRATION | 2
  DEPRESSED LEVEL OF CONSCIOUSNESS | 2

3. Secondary Outcome: Objective Response Rate
Description: Objective Response Rate (ORR) = CR+ PR. ORR is evaluated per RECIST v1.1 criteria.
  Complete Response (CR): Disappearance of all target lesions; Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions.
Time Frame: From start of study treatment until disease progression or death, whichever occurs first.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ENMD-2076
Number analyzed (Participants) | 25
percentage of participants | 8 [1 to 26]

ADVERSE EVENTS:
Arm/Group | ENMD-2076
Serious Adverse Events (participants affected / at risk) | 7/25
Other Adverse Events (participants affected / at risk) | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ENMD-2076 (N=25)
Agitation (Psychiatric disorders) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Colitis (Gastrointestinal disorders) | 1
Confusion (Psychiatric disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Depressed level of consciousness (Nervous system disorders) | 1
Diarrhea (Gastrointestinal disorders) | 2
Fatigue (General disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Edema limbs (General disorders) | 1
Lung infection (Infections and infestations) | 2
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ENMD-2076 (N=25)
HYPERTENSION (Vascular disorders) | 19
HYPOALBUMINEMIA (Metabolism and nutrition disorders) | 17
FATIGUE (General disorders) | 16
LYMPHOCYTE COUNT DECREASED (Investigations) | 14
NAUSEA (Gastrointestinal disorders) | 13
DIARRHEA (Gastrointestinal disorders) | 11
PROTEINURIA (Renal and urinary disorders) | 13
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 11
CONSTIPATION (Gastrointestinal disorders) | 12
PLATELET COUNT DECREASED (Investigations) | 11
DYSPEPSIA (Gastrointestinal disorders) | 11
DIZZINESS (Nervous system disorders) | 9
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 8
DRY MOUTH (Gastrointestinal disorders) | 8
HEADACHE (Nervous system disorders) | 8
GLUCOSE INTOLERANCE (Metabolism and nutrition disorders) | 7
HYPONATREMIA (Metabolism and nutrition disorders) | 6
INSOMNIA (Psychiatric disorders) | 7
ALKALINE PHOSPHATASE INCREASED (Investigations) | 7
MUCOSITIS ORAL (Gastrointestinal disorders) | 7
EDEMA LIMBS (General disorders) | 6
VOMITING (Gastrointestinal disorders) | 5
HEMATURIA (Renal and urinary disorders) | 6
ABDOMINAL PAIN (Gastrointestinal disorders) | 6
ANEMIA (Blood and lymphatic system disorders) | 6
ANXIETY (Psychiatric disorders) | 6
BACK PAIN (Musculoskeletal and connective tissue disorders) | 6
WHITE BLOOD CELL DECREASED (Investigations) | 6
ELECTROCARDIOGRAM QT CORRECTED INTERVAL (Cardiac disorders) | 5
NON-CARDIAC CHEST PAIN (General disorders) | 5
URINARY TRACT INFECTION (Renal and urinary disorders) | 5
CREATININE INCREASED (Investigations) | 4
FEVER (General disorders) | 4
HYPERURICEMIA (Metabolism and nutrition disorders) | 4
HYPOMAGNESEMIA (Metabolism and nutrition disorders) | 4
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 4
COUGH (Respiratory, thoracic and mediastinal disorders) | 4
ANOREXIA (Metabolism and nutrition disorders) | 4
BLOOD BILIRUBIN INCREASED (Investigations) | 4
ALOPECIA (Skin and subcutaneous tissue disorders) | 3
DYSGEUSIA (Nervous system disorders) | 3
FLATULENCE (Gastrointestinal disorders) | 3
FLU LIKE SYMPTOMS (General disorders) | 3
HOARSENESS (Respiratory, thoracic and mediastinal disorders) | 3
PALMAR-PLANTAR ERYTHRODYSESTHESIA SYNDRO (Skin and subcutaneous tissue disorders) | 3
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 3
SINUS TACHYCARDIA (Cardiac disorders) | 3
WEIGHT GAIN (Investigations) | 3
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 3
HYPERKALEMIA (Metabolism and nutrition disorders) | 2
NEUTROPHIL COUNT DECREASED (Investigations) | 3
HYPOGLYCEMIA (Metabolism and nutrition disorders) | 3
HYPOKALEMIA (Metabolism and nutrition disorders) | 3
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2
BLURRED VISION (Eye disorders) | 2
DRY SKIN (Skin and subcutaneous tissue disorders) | 2
DYSPHAGIA (Gastrointestinal disorders) | 2
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 2
HYPERTHYROIDISM (Endocrine disorders) | 2
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 2
PARESTHESIA (Nervous system disorders) | 2
SINUS BRADYCARDIA (Cardiac disorders) | 2
TOOTHACHE (Gastrointestinal disorders) | 2
URINARY FREQUENCY (Renal and urinary disorders) | 2
WEIGHT LOSS (Investigations) | 2
BONE PAIN (Musculoskeletal and connective tissue disorders) | 2
CONCENTRATION IMPAIRMENT (Nervous system disorders) | 2
HEMOGLOBIN INCREASED (Investigations) | 2
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 2
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 2
GGT INCREASED (Investigations) | 2
HYPOCALCEMIA (Metabolism and nutrition disorders) | 2
MYALGIA (Musculoskeletal and connective tissue disorders) | 2
DEPRESSION (Psychiatric disorders) | 2
EDEMA TRUNK (General disorders) | 2
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 2
LIPASE INCREASED (Investigations) | 2
GENERALIZED MUSCLE WEAKNESS (Musculoskeletal and connective tissue disorders) | 2
HYPOPHOSPHATEMIA (Metabolism and nutrition disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes